CLINICAL TRIAL: NCT04424095
Title: Investigation of Chronic Venous Disease in Pediatric Population
Brief Title: Venous Disease in Pediatric Population
Acronym: VEDIPEDI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Associate Professor of Vascular Surgery, University of Catanzaro
Other Study IDs: ER.ALL.2018.21
Record Dates: First submitted 2020-06-06; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Chronic Venous Insufficiency; Pediatric ALL
Keywords: Chronic venous disease; Pediatrics; vein reflux
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients: Recruited pediatric patients will undergo an in-office vascular visit and an echo duplex scan of lower limbs, in order to detect any symptoms or signs related to chronic venous disease.
  Interventions: Diagnostic Test: In-office vascular visit; Diagnostic Test: Echo Duplex of lower limbs

INTERVENTIONS:
Diagnostic Test: In-office vascular visit — The patient will be examined to search for signs or symptoms of chronic venous disease (teleangiectasia, reticular veins, varicose veins, skin changes, pain, itching, heavy legs, ankle edema)
Diagnostic Test: Echo Duplex of lower limbs — The venous system of lower limbs will be checked in order to detect any vein dilation and reflux.

SUMMARY:
Chronic venous disease (CVD) is widespread in adult subjects of western countries and is responsible of important morbidity and healthcare costs. CVD has never been extensively studied in pediatric population where the early pathophysiological alterations may occur undetected. The aim of this study is to assess the prevalence of CVD searching also for the early clinical and instrumental signs of this disease.

DETAILED DESCRIPTION:
Chronic venous disease (CVD) of lower limbs for its high prevalence in adult population represents one of the main causes of morbidity in western countries, and it has also an important effect on healthcare cost absorbing 1-2% of the total health budget in western countries. Clinical manifestations related to CVD are well documented in adults, with clinical guidelines that standardize both diagnosis and treatment. Nevertheless, there is a scarcity of published data regarding CVD in children, and in addition, venous duplex ultrasound test of the lower limbs is performed much less commonly in children than in adults.

Therefore, the natural history of pediatric venous reflux remains unclear, although it is possible that it precedes the onset of CVD in adulthood. In this context, this observational study aims to identify the presence of venous reflux, as well as clinical and morphological data in pediatric subjects, aged between 9 and 18 years old, by performing an office vascular visit and an echo duplex scan of lower limbs. The endpoints of this study are to prospectively assess the prevalence of CVD in children, as well as to evaluate a possible correlation between vein diameter and pathological vein reflux.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Patients

Exclusion Criteria:

* Patients with mental retardation
* Patients with Marfan syndrome
* Patients with an inability to stand or collaborate for the clinical tests.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric subjects, of both sex, aged between 9 and 18 years old which are cooperative for visit and diagnostic testing.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Chronic Venous Disease | at 9 month
  The Prevalence of Chronic Venous Disease in the population study will be assessed.
Echo duplex evaluation | at 10 month
  The correlation between veins diameter and the presence of reflux will be evaluated in pediatric population

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Serra, M.D., Ph.D., Principal Investigator — University Magna Graecia of Catanzaro
Locations (1):
- University Magna Graecia of Catanzaro, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robertson L, Evans C, Fowkes FG. Epidemiology of chronic venous disease. Phlebology. 2008;23(3):103-11. doi: 10.1258/phleb.2007.007061. PMID 18467617
- [Background] Beebe-Dimmer JL, Pfeifer JR, Engle JS, Schottenfeld D. The epidemiology of chronic venous insufficiency and varicose veins. Ann Epidemiol. 2005 Mar;15(3):175-84. doi: 10.1016/j.annepidem.2004.05.015. PMID 15723761
- [Background] Griffiths L, Vasudevan V, Myers A, Morganstern BA, Palmer LS. The role of inheritance in the development of adolescent varicoceles. Transl Androl Urol. 2018 Dec;7(6):920-925. doi: 10.21037/tau.2018.09.02. PMID 30505728